CLINICAL TRIAL: NCT00891722
Title: Translation Study for Children and Adolescents With Low Grade Glioma
Brief Title: Tumor Tissue, Blood Samples, and Family History in Predicting Tumor Development and Response to Treatment in Young Patients With Low-Grade Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000614912; CCLG-CNS-2007-13-TRANSCAL; EU-20879
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood brain stem glioma; untreated childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; untreated childhood cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood cerebral astrocytoma; childhood oligodendroglioma; recurrent childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway and hypothalamic glioma; childhood mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Optic Nerve Glioma

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand why low-grade gliomas develop in young patients and predict how they will respond to treatment.

PURPOSE: This clinical trial is studying tumor tissue, blood samples, and family history in predicting tumor development and response to treatment in young patients with low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop a better understanding of why low-grade glioma tumors develop in children and adolescents.
* To study genetic profiles that may predict response to treatment and provide clues to how these tumors developed initially using tumor and blood samples from these patients.

OUTLINE: This is a multicenter study.

* Retrospective data collection (for participants recruited from study SIOP-LGG1): During a follow-up appointment for study SIOP-LGG1, both biological parents* are asked to complete a questionnaire about their family's cancer history. They may complete the questionnaire either in the clinic or in their home. Participants may complete and return the questionnaires at any time throughout the study.
* Prospective data collection (for participants recruited from study SIOP-LGG-2004): Both biological parents* are asked to complete a family history questionnaire and provide information about their family's cancer history. Participants may complete and return the questionnaires at any time throughout the study.

NOTE: *In circumstances where either or both biological parents are unable to complete the questionnaire, it may be completed by the patient diagnosed with low grade glioma (if they are over 16 years old) or adoptive parents or guardians, if they feel they have the knowledge to complete the questionnaire.

Tumor tissue and blood samples collected on SIOP-LGG1 or SIOP-LGG-2004 are analyzed for genetic profiles predictive of response to treatment and for different patterns of tumor development, natural tumor behavior, and tumor sensitivity to cancer therapies. Collected family data are anonymised and linked to the biological sample collected. Samples are then stored for future molecular genetic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biological parents of a child or adolescent patient diagnosed with low grade glioma (LGG)

  * LGG patients participating in 1 of the following clinical trials:

    * On active follow up for study SIOP-LGG1 at a Children's Cancer and Leukemia Group center
    * On study SIOP-LGG-2004
  * Adoptive parents or guardians allowed if they feel they have the knowledge to complete the study questionnaire, provided either or both biological parents are unable to complete the questionnaire

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
Identification of factors that could determine different patterns of tumor development, natural tumor behavior, and tumor sensitivity to therapies

CONTACTS AND LOCATIONS:
Overall Officials: David A. Walker, Principal Investigator — Queen's Medical Center
Locations (1):
- Queen's Medical Centre, Nottingham, England, United Kingdom